CLINICAL TRIAL: NCT00350857
Title: A Phase IV, Multi-Center, Open-Label, Safety and Effectiveness Study of Extended-Release Carbamazepine in the Treatment of Mania in Children and Adolescents Aged 10-17 Years With Acute Manic or Mixed Bipolar I Disorder.
Brief Title: The Young Adult and Pediatric Bipolar Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Validus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD417-311
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2009-11

CONDITIONS: Bipolar I Disorder

ARMS (1):
- Equetro active (Active Comparator)
  Interventions: Drug: Extended-Release Carbamazepine

INTERVENTIONS:
Drug: Extended-Release Carbamazepine

SUMMARY:
To examine the safety and effectiveness of extended-release carbamazepine in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Key Inclusion Criteria:

  1. DSM-IV diagnosis of bipolar I disorder, most recent episode manic or mixed.
  2. A lifetime history of bipolar disorder symptoms for at least 2 months.
  3. YMRS score greater than or equal to 16.
  4. CGI-S score greater than or equal to 4.
  5. Male or female outpatient aged between 10-17 years old inclusive at the time of consent.
  6. Functioning at an age-appropriate level intellectually, as deemed by the Investigator.
  7. The subject has no co-morbid illness that could affect efficacy, safety, or tolerability or in any way interfere with the subject's participation in the study.
  8. Must have a satisfactory medical assessment with no clinically significant and relevant abnormalities.

Exclusion Criteria:

* Key Exclusion Criteria:

  1. Current controlled or uncontrolled, co-morbid psychiatric diagnosis that could interfere with clinical assessments or study conduct.
  2. A history of lack of therapeutic response or hypersensitivity to the study drug.
  3. A greater than or equal to 50% reduction in YMRS between Screening and Baseline.
  4. Acutely at risk for suicidal or violent behavior or a history of suicide attempts requiring medical intervention.
  5. A history of aplastic anemia, agranulocytosis or bone marrow depression.
  6. A history of seizure disorder, other than a single childhood febrile seizure.
  7. A history of severe, unstable asthma.
  8. Current hospitalization for psychiatric symptoms.
  9. History of alcohol or other substance abuse or dependence.
  10. Pregnant or lactating females.
  11. Body weight less than or equal to 25 kg.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by the occurrence of treatment emergent adverse events and evaluations of clinical laboratory values, physical examinations, vital signs and ECG data after 6 months of treatment. | 6 months

SECONDARY OUTCOMES:
Reduction of bipolar symptoms as assessed by the Young Mania Rating Scale (YMRS), Clinical Global Impressions Scale (CGI) and Children's Depression Rating Scale (CDRS-S) after 6 months of treatment. | 6 months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - 11 Shire Clinical Research Site, Altamonte Springs, Florida
  - 17 Segal Institute for Clinical Research, Fort Lauderdale, Florida
  - 19 Sarkis Clinical Trials, Gainesville, Florida
  - 23 Shire Clinical Research Site, Jacksonville, Florida
  - 21 Scientific Clinical Research, North Miami, Florida
  - 14 Northlake Medical Research, Decatur, Georgia
  - 04 Mountain West Clinical Trials, Eagle, Idaho
  - 25 Capstone Clinical Research, Libertyville, Illinois
  - 15 Psychiatric Associates, Overland Park, Kansas
  - 27 Owensboro Behavioral Care, Owensboro, Kentucky
  - 05 Brentwood Research Institute, Shreveport, Louisiana
  - 13 Pharmasite Research, Inc, Baltimore, Maryland
  - 02 Finger Lakes Clinical Research, Rochester, New York
  - 01 Nccacrf, Chapel Hill, North Carolina
  - 06 University of Cincinnati, College of Medicine, Cincinnati, Ohio
  - 09 Discovery and Wellness Center for Children, Cleveland, Ohio
  - 03 IPS Research, Oklahoma City, Oklahoma
  - 26 Suburban Research Associates, Media, Pennsylvania
  - 12 Claghorn-Lesem Research Clinic, Bellaire, Texas
  - 07 Center for Pediatric Psychiatry, Dallas, Texas
  - 24 Red Oak Psychiatry Associates, Houston, Texas
  - 10 RID Clinical Research, Inc, Lake Jackson, Texas
  - 08 Dominion Clinical Research, Midlothian, Virginia
  - 22 Brighton Research Group, Virginia Beach, Virginia
  - 20 Shire Clinical Research Site, Milwaukee, Wisconsin
  - 16 Rogers Center for Research and Training, Milwaukee, Wisconsin